CLINICAL TRIAL: NCT07053306
Title: Protocol III: SGLT2i, Ketoacidosis, Volume Contraction, and Insulinopenia
Brief Title: SGLT2i, Ketoacidosis, Volume Contraction, and Insulinopenia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20230457HU - 504076; R01DK024092 (NIH)
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
Keywords: Pancreatic clamp; Endogenous glucose production; Ketogenesis; Gluconeogenesis; Lipolysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: A randomized controlled 1 arm clinical trial comprised of 4 studies
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin (Experimental): Empagliflozin 25 mg/day
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — A medication used in the management and treatment of type 2 diabetes mellitus. It is in the sodium-glucose co-transporter (SGLT-2) class of medications.
  Other Names: Jardiance

SUMMARY:
To examine the 2-HIT hypothesis that the SGLT2i-induced stimulation of EGP, lipolysis, and ketone production requires the combination of volume depletion plus insulinopenia in T2D individuals.

DETAILED DESCRIPTION:
After screening visit, subjects will participate in four additional visits and or at least one of the four visits that will be performed in random order starting at 6:00 AM to the Clinical Research Center at University Hospital-Texas Diabetes Institute.

Visit 2 (Study 1): At 6:00AM at (Study 1), a prime-continuous infusions of 6,6, D2-Glucose or U-3H-glucose and U-2H-glycerol or U-14C-Glycerol are started and continued to study end (2:00 PM) to measure rates of hepatic glucose production (HGP) and fat break down (lipolysis).3H-Glucose infusion to be given: (Prime=25µCi x (FPG/100), Continuous=0.25µCi/min x 480 min=120µCi). At time zero (9:00 AM) subjects will ingest Empagliflozin (25 mg). Plasma substrate, hormone concentrations, U-3H-glucose and U-14C-glycerol specific activities will be measured every 5-30 minutes for 300 minutes (2:00 PM) and 295 minutes. If Principal Investigator (PI) use U-2H-glycerol instead of U-14C Glycerol, PI will measure plasma U-2H-glycerol enrichment instead of U-14C-glycerol specific activities. Detailed explanation on page 54, if PI will use U-6,6, D2-Glucose instead of U-3H Glucose, PI will measure plasma 2H-Glucose enrichment instead of 3H Glucose specific activities. Detailed explanation on page 54.

Visit 3 (Study 2, Optional): At 6:00AM prime-continuous infusions of 6,6, D2-Glucose or U-3H-Glucose and U-2H-glycerol or U-14C-Glycerol are started and continued to study end (2:00 PM) to measure rates of hepatic glucose production (HGP) and lipolysis. 3H-Glucose infusion to be given: (Prime=25µCi x (FPG/100), Continuous=0.25µCi/min x 480 min=120µCi). At 7 AM an infusion of normal saline will be started at the rate of 150 ml/hour and continued to the end of study at 2 PM (total volume = 1050 ml; total Na and Cl = 154 meq) to provide volume replacement for blood loss. At time zero (9:00 AM) subjects will ingest Empagliflozin (25 mg). Plasma substrate, hormone concentrations, 3H-glucose and 14C-glycerol specific activities will be measured every 5-30 minutes for 300 minutes (2:00 PM) and 295 minute. If PI use U-2H-glycerol instead of U-14C Glycerol, PI will measure plasma U-2H-glycerol enrichment instead of U-14C-glycerol specific activities. Detailed explanation on page 55. If PI use U-6,6, D2-Glucose instead of U-3H Glucose, PI will measure plasma 2H-Glucose enrichment instead of 3H Glucose specific activities. Detailed explanation on page 55.

Visit 4 (Study 3, Optional): At 6:00AM prime-continuous infusions 6,6, D2-Glucose or U-3H-Glucose and U-2H-glycerol or U-14C-Glycerol are started and continued to study end (2:00 PM) to measure rates of Hepatic Glucose Production (HGP) and fat break down (lipolysis). 3H-Glucose infusion to be given: (Prime=25µCi x (FPG/100), Continuous=0.25µCi/min x 480 min=120µCi). At time zero (9:00 AM) subjects will ingest Empagliflozin (25 mg) and octreotide or somatostatin with insulin and glucagon will be given to reduce volume without insulinopenia. Plasma substrate and hormone concentrations and 3H-glucose/14C-glycerol specific activities will be measured every 5-30 minutes for 300 minutes (2:00 PM) and 295 minute. If PI use U-2H-glycerol instead of U-14C Glycerol, PI will measure plasma U-2H-glycerol enrichment instead of U-14C-glycerol specific activities. Detailed explanation on page 55-56. If PI uses U-6,6, D2-Glucose instead of U-3H Glucose, PI will measure plasma 2H-Glucose enrichment instead of 3H Glucose specific activities. Detailed explanation on page 56.

Visit 5 (Study 4, Optional): At 6:00AM prime-continuous infusions of 6,6, D2-Glucose or 3H-Glucose and U-2H-glycerol or U-14C-Glycerol are started and continued to study end (2:00 PM) to measure rates of hepatic (liver) glucose production (HGP) and fat break down (lipolysis). 3H-Glucose infusion to be given: (Prime=25µCi x (FPG/100), Continuous=0.25µCi/min x 480 min=120µCi). At 7 AM an infusion of normal saline will be started at the rate of 150 ml/hour and continued to the end of study at 2 PM (total volume = 1050 ml; total Na and Cl = 154 meq) to provide volume replacement for blood loss. At time zero (9:00 AM) subjects will ingest empagliflozin (25 mg) and octreotide or somatostatin with insulin and glucagon will be given. Plasma substrate and hormone concentrations and 3H-glucose/14C-glycerol specific activities will be measured every 5-30 minutes for 300 minutes (2:00 PM) and 295 minute. If PI uses U-2H-glycerol instead of U-14C Glycerol, PI will measure plasma U-2H-glycerol enrichment instead of U-14C-glycerol specific activities. Detailed explanation on page 56. If PI use U-6,6, D2-Glucose instead of U-3H Glucose, PI will measure plasma 2H-Glucose enrichment instead of 3H Glucose specific activities. Detailed explanation on page 56.

In Substudy II, PI will use stable isotopes (6,6-D2-glucose and U-2H-glycerol) or radioisotopes (U-3H-glucose and U-14C-glycerol) to measure endogenous glucose production (EGP) and fat breakdown (lipolysis), depending on isotope availability and cost. Both sets of isotopes will provide the necessary data to address research objectives.

ELIGIBILITY:
Patients with T2D

Inclusion Criteria:

* Ages 30-75 years
* Body Mass Index (BMI) 21-45 kg/m2
* Hemoglobin A1C (HbA1c) = 7.0-11%
* Estimated glomerular filtration rate (eGFR) > 60 ml/min/1.73m2
* Blood Pressure (BP) < 160/90 mmHg
* Participants must be in general good health based on medical history, physical exam, screening blood chemistries, complete blood chemistry (CBC), thyroid stimulating hormone/thyroxine (TSH/T4), electrocardiogram (EKG), and urinalysis
* Stable body weight (±1.5 kg) over the last 3 months and must not participate in an excessively heavy exercise program
* Patients treated with diet, sulfonylurea (SU), metformin (MET), or SU/MET
* Statin therapy is permissible if the dose has been stable for at least 3 months

Exclusion Criteria:

* Patients treated with Glucagon-like peptide 1 receptor agonists (GLP-1 RA), Dipeptidyl Peptidase IV inhibitors (DPP-4i), Thiazolidinediones (TZD), or insulin are excluded
* Patients taking medications (other than SU/MET) known to affect glucose metabolism are excluded
* Subjects with evidence of proliferative retinopathy or eGFR < 60 are excluded
* Women of childbearing potential are excluded unless they are taking/using appropriate contractive medications/devices

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Ketone Body Turnover (ketogenesis) | 0 and 300 minutes
  Measurement of ketone body turnover rate during the baseline state and 240-300-minute time period, before and after Empagliflozin administration.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph DeFronzo, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Texas Diabetes Institute/UH, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with NIH and as a publication in a peer reviewed journal once data are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At study end after analysis of data.